CLINICAL TRIAL: NCT04191343
Title: A Single-arm, Single-center, Prospective Clinical Study on the First-line Treatment of Advanced Biliary System Tumors With Tripley Monoclonal Antibody Combined With GEMOX Regimen
Brief Title: Clinical Study on the First-line Treatment of Advanced Biliary System Tumors With Tripley Monoclonal Antibody Combined With GEMOX Regimen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2019-91
Record Dates: First submitted 2019-12-06; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Advanced Biliary Tract Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The control group (Experimental)
  Interventions: Drug: Toripalimab injection combined with GEMOX

INTERVENTIONS:
Drug: Toripalimab injection combined with GEMOX — Toripalimab Injection (240mg, intravenous drip, d1, q3w);Combined with gemcitabine (1000mg/m2, intravenous drip, d1, d8, q3w) and oxaliplatin (100mg/m2, intravenous drip, d1, q3w)

SUMMARY:
This is an open, single-arm, single-center, prospective phase II clinical study to evaluate the efficacy and safety of first-line tripletrumab combined with GEMOX chemotherapy in patients with advanced biliary tract tumors.

Selected patients will receive the following treatment:

Triplel monoclonal antibody (240mg, intravenous drip, d1, q3w);Combined with gemcitabine (1000mg/m2, intravenous drip, d1, d8, q3w) and oxaliplatin (100mg/m2, intravenous drip, d1, q3w) until the disease progresses or an intolerable adverse reaction occurs (the maximum treatment time is 2 years).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75.
* KPS score ≥80 points within 7 days before inclusion.
* For subjects with previously untreated advanced or metastatic biliary tract systemic tumors (gallbladder cancer, intrahepatic and extrahepatic cholangiocarcinoma), or who have previously undergone radical surgery + adjuvant therapy, the metastatic lesions should be detected for the first time at ≥6 months after the last adjuvant treatment, and the pathological type is adenocarcinoma.
* In CT/MRI examination, there was at least one measurable lesion according to RECIST1.1 criteria.
* The blood routine and biochemical indicators of the subject within 7 days before enrollment meet the following standards:

  1. Hemoglobin ≥90g/L; Absolute count of neutrophils (ANC) ≥1.5×109/L; Platelet ≥100×109/L (patients should not receive blood transfusion or growth factor support within 14 days after blood collection);
  2. ALT and AST≤2.5 times normal upper limit (ULN); ALP 2.5 x ULN or less;
  3. Total bilirubin <1.5 ULN (patients with Gilbert syndrome can be included if total bilirubin <3 ULN);
  4. Serum creatinine <1.5 ULN or estimated glomerular filtration rate ≥60ml/min/1.73m2 (appendix 3);
  5. Serum albumin≥30g/L;
  6. International standardized ratio (INR) or prothrombin time (PT) ≤1.5 ULN, unless the patient is receiving anticoagulant therapy and PT is within the anticoagulant expected treatment range;
  7. Activated partial thromboplastin time (APTT) ≤1.5 times ULN.
* Be able to follow the protocol during the study period. 7) provide written informed consent before entering the study, and patients have been informed that they can withdraw from the study at any time without any loss.
* Fertile women (appendix 6) must test negative for urine or serum pregnancy within 7 days prior to enrollment and must agree to use effective contraception for at least 120 days during the study period and after the last administration (including chemotherapy and triplegizumab).
* Unsterilized men must agree to use effective contraception during the study period and for at least 120 days after their last dose.

Exclusion Criteria:

* Previous treatment for biliary tract tumors, including radiotherapy, chemotherapy and immunotherapy (except for patients with recurrence more than 6 months after the end of previous adjuvant therapy)
* Patients with active autoimmune diseases or a history of autoimmune diseases that may recur . Note: patients with the following diseases are not excluded and can be further screened:

  1. controlled type 1 diabetes
  2. hypothyroidism (which can be controlled with hormone replacement therapy alone)
  3. controlled celiac disease
  4. skin diseases that require no systemic treatment (e.g. Vitiligo, psoriasis, alopecia)
  5. Any other disease that is not expected to recur in the absence of an external trigger
* Any active malignancy within 2 years, except for specific cancers being studied in this trial and locally recurrent cancers that have been cured (such as excised basal or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ).
* There was uncontrollable pleural effusion, pericardial effusion or ascites requiring frequent drainage within 14 days prior to enrollment (cytological examination of effusion was allowed).
* Patients with gastrointestinal bleeding within the first two weeks of inclusion, or those with high blood risk as judged by the researchers.
* Gastrointestinal perforation and/or fistula occurred within 6 months before admission.
* Body weight loss≥20% in the first 2 months.
* Lung diseases of clinical significance: interstitial pulmonary disease, non-infectious pneumonia, pulmonary fibrosis, acute pulmonary disease, etc.
* Uncontrollable systemic diseases including diabetes, hypertension, etc.
* Severe chronic or active infections, including tuberculosis and HIV infection, that require systemic antibacterial, antifungal or antiviral treatment.
* Untreated chronic hepatitis b or chronic HBV carriers with hepatitis b virus (HBV) DNA exceeding 1000 IU/mL, or hepatitis c virus (HCV) RNA positive patients should be excluded. Nonactive hepatitis b surface resistance Original (HBsAg) carriers, treated and stable hepatitis b patients (HBV DNA <1000IU/mL), and cured hepatitis c patients may be included.
* Any of the following cardiovascular risk factors:

  1. The occurrence of cardiogenic chest pain within no more than 28 days before enrollment was defined as moderate pain with limited daily living activities.
  2. Symptomatic pulmonary embolism occurred within 28 days or less before enrollment.
  3. Acute myocardial infarction occurred within less than 6 months before inclusion.
  4. Any history of heart failure reaching the New York heart association level III/IV (appendix 5) less than 6 months prior to enrollment.
  5. Ventricular arrhythmias of grade 2 or greater occurred within less than 6 months before inclusion, or were accompanied by supraventricular tachyarrhythmias requiring drug treatment.
  6. Cerebrovascular accident (CVA) occurred within less than 6 months before inclusion.
* Peripheral nerve disease is known to exceed NCI-CTCAE level 1. CTCAE 1However, patients with only deep tendon reflex (DTR) disappearance need not be excluded.
* Moderate or severe renal impairment [creatinine resolution equal to or less than 50 ml/min (based on the Cockroft and Gault equations)], or serum creatinine > normal upper limit (ULN).
* Allergic to any component of the study drug.
* Have undergone allogeneic stem cell transplantation or organ transplantation.
* Corticosteroids (prednisone with a dose higher than 10 mg/d or similar drugs) should be used within 14 days before enrollment Isodose) or other immunosuppressant systemic therapy. Note: patients who currently or previously used any of the following steroid regimens may be included:

  1. Adrenalin alternative steroids (prednisone≤10mg/d or equivalent)
  2. Topical, intraocular, intraarticular, intranasal and inhaled corticosteroids with minimal systemic absorption.
  3. Short-term (≤7 days) use of corticosteroids for prophylaxis (e.g Antiemetic agents for specific chemotherapy) or for the treatment of non-autoimmune conditions (such as delayed hypersensitivity caused by exposure to allergens).
* Received live vaccine within 4 weeks prior to enrollment. (note: seasonal influenza vaccines are usually inactivated vaccines and are permitted. Vaccines used in the nasal cavity are live vaccines and should not be used.
* Received: immunotherapy within 28 days prior to enrollment or within 5 half-lives (whichever is shorter, but at least 14 days) Treatment (such as interleukin, interferon, thymosin, etc.) or any experimental treatment.
* Palliative radiotherapy was given within 14 days prior to enrollment.
* Have received anti-pd-1, anti-pd-l1, anti-pd-l2 or any other specific targeted t-cell co-stimulation or checkpoint pathway antibody or drug therapy.
* Receive major surgery within 28 days prior to enrollment, unless the surgery is minimally invasive (e.g., central venous catheterization through peripheral venipuncture [PICC]).
* In the case of uncontrolled epilepsy, CNS disease or mental disorder, the investigator shall determine whether the clinical severity interferes with the signing of the informed consent or affects the patient's oral medication compliance.
* There are potential medical conditions or alcohol/drug abuse or dependence that researchers consider to be detrimental to the study of drug administration or to the interpretation of drug toxicity or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 2 years
  Objective response rate (ORR) on imaging of Toripalimab combined with chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Haijun Zhong, Zhenjiang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided